CLINICAL TRIAL: NCT05731284
Title: Platelet Rich Plasma as an Adjunct Therapy at the Time of Transvaginal Native Tissue Prolapse Surgery
Acronym: PRP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Isuzu Meyer, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-300009943
Record Dates: First submitted 2023-01-26; First posted 2023-02-16 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Masking: Participants and study examiners performing the postoperative assessment will remain masked to the intervention assignment for the study duration, unless a medical indication for unmasking is identified.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adjunct Platelet rich plasma (PRP) therapy (Active Comparator): Study Interventions: PRP will be injected in a systematic grid like fashion into the fibromuscular connective tissue of the anterior compartment following vaginal incision and dissection.
  Interventions: Procedure: Platelet rich plasma (PRP) Injection
- Normal saline (Placebo Comparator): Placebo: Normal saline will be injected in a systematic grid like fashion into the fibromuscular connective tissue of the anterior compartment following vaginal incision and dissection.
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Platelet rich plasma (PRP) Injection — Randomly picked (like the flip of a coin) by a computer to receive either platelet-rich plasma (PRP) or normal saline. This is a double-blind study. During vaginal prolapse surgery, the surgeon will inject PRP into the vaginal tissue at the surgical site.
  Arms: Adjunct Platelet rich plasma (PRP) therapy
Procedure: Placebo — Normal saline Injection
  Arms: Normal saline

SUMMARY:
The purpose of the study is to evaluate the surgical outcomes of injecting platelet-rich plasma (PRP) into the vaginal tissue as an adjunct therapy at the time of prolapse surgery

DETAILED DESCRIPTION:
Platelet rich plasma (PRP) is an autologous product with high levels of platelets which are concentrated with bioactive growth factors responsible for accelerating tissue healing by stimulating the number of reparative cells to create collagen production, angiogenesis and neurogenesis. The overarching goal is to evaluate the effectiveness and safety of the adjunct application of PRP in the fibromuscular connective tissue (the site of anterior tissue plication) at the time of anterior colporrhaphy (the site of highest recurrence risk) in women undergoing native tissue vaginal prolapse repair, to promote tissue healing and regeneration, thus to improve surgical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Desire surgical treatment via a transvaginal native tissue approach.
* Completed child-bearing

Exclusion Criteria:

* Unable to follow-up, not willing to, or unable to participate in the proposed study
* Prior pelvic surgery within the past 12 months
* Prior anterior/apical suspension procedures
* Prior graft augmented prolapse surgery
* Pelvic/abdominal radiation
* Pelvic mass
* History of solid organ malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Anterior wall descensus measured by the POP-Q System, Ba point | 12 month
  Anterior wall descensus measured by the POP-Q System, Ba point

SECONDARY OUTCOMES:
Apical wall descensus measured by the POP-Q System, C point | 12 months
  Apical wall descensus measured by the POP-Q System, C point
Posterior wall descensus | 12 months
  Posterior wall descensus measured by the POP-Q System, Bp point
Leading edge | 12 months
  leading edge (Ba, C, or Bp) beyond the hymen (>0)
Safety outcomes | 12 months
  operative time, blood loss, intra-, peri/postoperative adverse events
Subjective | 12 months
  Bothersome vaginal bulge symptoms (positive response to "usually have a bulge or something falling out that you can see or feel in your vaginal area" from the PFDI-20)
Retreatment | 12 months
  Retreatment for prolapse: pessary or surgery - dichotomous (failure: retreatment)

CONTACTS AND LOCATIONS:
Overall Officials: Isuzu Meyer, MD, MSPH, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No